CLINICAL TRIAL: NCT02987738
Title: A Randomized, Double-Blind, Placebo-controlled, Single-center, Phase 1 Inpatient Pilot Study to Explore the Safety and Efficacy of DAPAglifozin as Add-on to Day and Night Closed-loop Control in Patients Type 1 Diabetes (T1D)
Brief Title: Pilot Study to Explore the Efficacy of DAPAglifozin as add-on to Closed-loop Control in Patients With Type 1 Diabetes
Acronym: DapaDream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Collaborators: AstraZeneca (Industry); Alcedis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ESR-15-11453
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Type1diabetes
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dapagliflozin (Experimental): two administrations of 10 mg dapagliflozin as tablet
  Interventions: Drug: Dapagliflozin
- Placebo Oral Tablets (Placebo Comparator): two administrations identical to the experimental drug
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin — two administrations in the evening and 12 hours later
  Other Names: Forxiga
  Arms: dapagliflozin
Drug: Placebo Oral Tablet — two administrations in the evening and 12 hours later
  Other Names: Control
  Arms: Placebo Oral Tablets

SUMMARY:
Dapagliflozin has a unique mechanism of action that does not directly affect either insulin resistance or insulin secretion, but rather improves glycemia by reduction of glucose re-absorption from proximal renal tubules. Dapagliflozin is expected to reduce mean daily glucose, improve glycemic control and reduce overall insulin requirements. Improved glycemic control with reduced variability may also lead to reduced frequency of hypoglycemia.

In youth with T1D, Dapagliflozin led to a significant reduction of insulin needed to achieve target glucose irrespective of preexisting HbA1c levels.

In this pilot study data will be collected to investigate the effect on glucose of two doses of 10mg (each) dapagliflozin within range for the ensuing 24 hours during the DreaMed automated insulin delivery in patients with type 1 diabetes dosing with dapagliflozin in an in-patient setting combined with an automated sensor based CE marked insulin delivery system to data if dapagliflozin is a suitable add-on therapy. This will provide optimal monitoring of subject safety and assessment of the effects of dapagliflozin in a structured setting.

If this inpatient study shows evidence that Dapagliflozin is a suitable add on therapy and leads to an increase of time within the target glucose range when using a sensor based insulin pump therapy (closed-loop) further outpatient studies are planned to be conducted.

DETAILED DESCRIPTION:
The purpose of this pilot study is to collect clinical data of two doses of 10mg (each) dapagliflozin as add-on to night and day closed-loop control using the DreaMed automated insulin delivery on the time [%] within glucose range 70-180 mg/dl (3.9-10mmol/l) for the ensuing 24 hours with two oral mixed-meals.

The study aimed to patients who have different degrees of inadequate glycemic control despite insulin use.

A maximum of 45 patients will be screened until 30 Type 1 Diabetes mellitus patient (15 adults, 15 adolescents) will completed the study.

The trial will consist of six visits: a screening visit (Visit 1), two dosing visits (Visit 2 and Visit 4), two phone visits (Visit 3 and Visit 5) and a follow-up visit (Visit 6). Furthermore, an information visit will take place prior to the screening visit in order to obtain patient's informed consent. Screening will take place 2-21 days prior to Visit 2 and the follow-up visit will take place 5-21 days after the end of Visit 4. The dosing visits will be separated by a wash-out period (5-30 days between the end of Visit 2 and begin of Visit 4) during which the subjects will resume their normal insulin treatment. Each phone visit (Visit 3 and Visit 5) will take place 3-5 days after the end of dosing Visits 2 and 4. The planned total duration of the trial is 18-78 days per subject (rescheduled visits excluded). Each subject will be randomised to a treatment sequence consisting of two treatment periods in which the subjects will receive 2 times 10mg dapagliflozin and placebo on two separate dosing visits.

Subjects metabolic control will be achieved by using the DreaMed system (closed loop). The procedure will be used in order to aim and maintain blood glucose levels between 70 and 180 mg/dl thereby.

Two standardized mixed-meals will be given 12 hours and 18 hours after dosing. Blood glucose measurements will be performed every 30min for 120min after the mixed-meal.

Blood samples for determination of dapagliflozin concentration in serum will be taken 14times in 24hours as well as ß-Hydroxybutyrate and every urine sample will be collected for 24 hours after first dosing for the determination of 24hour urinary glucose and creatinine for efficacy measurement.

In addition a full blood gas analysis will be drawn if an elevated β-hydroxybutyrate of >1.0 mmol/L will be detected.

24 hours after first dosing with dapagliflozin/ placebo of each dosing visit the subjects will resume their usual insulin treatment and can leave the hospital.

After conclusion of the trial the documented insulin doses over time will be summed up for calculation of the total insulin dose and the insulin dose per kg body weight per 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 12-21 years (both inclusive)
2. Type 1 diabetes mellitus (as diagnosed clinically) ≥ 12 months
3. No DKA 12 weeks prior to the study
4. On CSII (insulin pump therapy) since at least 3 months
5. Average daily dose of Insulin between 0.6 - 2.0 U/kg
6. Body mass index 18 to 35 kg/m2 or the 10th to 99th centile for BMI according to age and gender with a minimum weight of 50kg
7. A1c range 6,5% - 11% (inclusive)

Exclusion Criteria:

1. History of drug or alcohol abuse within the last five years prior to screening
2. Anamnestic history of hypersensitivity to the study drugs (or any component of the study drug) or to drugs with similar chemical structures
3. History of severe or multiple allergies
4. Treatment with any other investigational drug within 3 months prior to screening
5. Progressive fatal disease
6. History of significant cardiovascular, respiratory, gastrointestinal, hepatic (ALAT and/or ASAT > 3 times the normal reference range), renal (creatinine > 1.1 mg/dl in women and > 1.5 mg/dl in men), neurological, psychiatric and/or hematological disease as judged by the investigator
7. Pregnant or lactating women
8. Sexually active women of childbearing potential not consistently and correctly practicing birth control by implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomized partner
9. Lack of compliance or other similar reason that, according to investigator, precludes satisfactory participation in the study

   Target Disease Exclusions
10. History of Type 2 diabetes, maturity onset diabetes of young (MODY), pancreatic surgery or chronic pancreatitis
11. Any use of oral hypoglycemic agents within 12 months prior to the screening visit
12. History of diabetes ketoacidosis (DKA) within 12 weeks prior to prior to the screening visit
13. History of diabetes insipidus
14. History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 3 months prior to prior to the screening visit
15. Frequent episodes of hypoglycemia as defined by more than one episode requiring assistance, emergency care (paramedics or emergency room care) or glucagon therapy, or more than 2 unexplained episodes of symptomatic hypoglycemia within 3 months prior to the screening visit. An unexplained event is defined as an event that cannot be explained by circumstances such as dietary (e.g. missed meal), strenuous exercise, error in insulin dosing, etc.
16. Hypoglycemic unawareness
17. History of Addison's disease or chronic adrenal insufficiency

    Physical and Laboratory Test Findings
18. Aspartate aminotransferase (AST) > 2x Upper limit of normal (ULN)
19. Alanine aminotransferase (ALT) > 2x ULN
20. Serum total bilirubin > 2x ULN
21. Estimated GFR (eGFR) by the Modification of Diet in Renal Disease (MDRD) formula ≤ 60 ml/min/1.73m2. The renal function, eGFR will be estimated by the abbreviated MDRD, using laboratory measurements of serum creatinine collected at screening [eGFR (ml/min/1.73m2) = 175 x (standardized Scr)-1.154 x (Age)-0.203 x (0.742 if female) x (1.212 if Black)].
22. Hemoglobin ≤ 11.0 g/dl (110 g/l) for boys / men; hemoglobin ≤10.0 g/dl (100 g/L) for girls / women.
23. Creatine kinase (CK) > 3x ULN
24. Positive for hepatitis B surface antigen or anti-hepatitis C virus antibody.
25. Abnormal Free T4 Note: abnormal TSH value at screening will be further evaluated for free T4. Subjects with abnormal free T4 values will be excluded. A one-time retest may be allowed, as determined by the Investigator, after a minimum of 6 weeks following the adjustment of thyroid hormone replacement therapy in subject who have had a prior diagnosis of a thyroid disorder and who are currently receiving thyroid replacement therapy. Such cases should be discussed with the Investigator prior to retesting. The subject must have all screening procedures and laboratory assessments performed as part of this re-test, and all of these must meet enrolment eligibility criteria. The subject's number will, however, remain the same as initially assigned.

    Allergies and Adverse Drug Reaction
26. Allergies or contraindication to the contents of dapagliflozin tablets or insulin
27. Renal, Hepatic, Hematological/Oncological Diseases/Conditions
28. History of unstable or rapidly progressing renal disease
29. Conditions of congenital renal glucosuria
30. Renal allograft
31. Significant hepatic disease, including but not limited to, chronic active hepatitis and/or severe hepatic insufficiency
32. Documented history of hepatotoxicity with any medication
33. Documented history of severe hepatobiliary disease
34. History of hemoglobinopathy, with the exception of sickle cell trait (SA) or
35. thalassemia minor; or chronic or recurrent hemolysis
36. Donation of blood or blood products to a blood bank, blood transfusion, or
37. participation in a clinical study requiring withdrawal of > 400 mL of blood during the 6 weeks prior to the enrolment visit
38. Known immunocompromised status, including but not limited to, individuals who have
39. undergone organ transplantation or who are positive for the human immunodeficiency virus
40. Malignancy within 5 years of the screening visit (with the exception of treated basal cell or treated squamous cell carcinoma of the skin) Other Exclusion Criteria
41. Prisoners or subjects who are involuntarily incarcerated
42. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
43. Replacement or chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid taken for > 4 weeks within 3 months prior to Day -3 visit.

    NOTE: Topical or inhaled corticosteroids are allowed.
44. Any unstable endocrine, psychiatric, rheumatic disorders as judged by the Investigator.
45. Subject is, in the judgment of the Investigator, unlikely to comply with the protocol or has any severe concurrent medical or psychological condition that may affect the interpretation of efficacy or safety data.
46. Subject with any condition which, in the judgment of the Investigator, may render the subject unable to complete the study or which may pose a significant risk to the subject.
47. Subject is currently abusing alcohol or other drugs or has done so within the last 6 months.
48. Subject is a participating investigator, study coordinator, employee of an investigator or immediate family member of any of the aforementioned.
49. Administration of any other investigational drug within 30 days of planned enrolment to this study.
50. No clinical conditions or clinically significant abnormalities, in any laboratory value(s) collected after screening and prior to randomization which, in the Investigator's judgment, should preclude entry into the treatment period.

    Dosing day exclusion criteria
51. Subjects who meet one or more of the dosing day exclusion criteria will be excluded from the dosing visit or withdrawn from the trial as specified below:
52. Non-fasting, ie, consumption of food or beverages other than water, later than at 23:00 hours the evening before dosing.
53. Clinically significant illness with onset within 4 weeks prior to dosing
54. Presence of clinically significant acute gastrointestinal symptoms (eg nausea, vomiting, heartburn or diarrhoea), as judged by the investigator
55. Consumption of alcohol within 24 hours prior to dosing
56. Episode of severe hypoglycemia occurring within the last 24 hours prior to dosing
57. Any medical condition that, in the opinion of the Investigator, could interfere with insulin pharmacokinetics and/or glucose metabolism.
58. Use of the following: systemic (oral or i.v.) corticosteroids, monoamine oxidase (MAO) inhibitors, systemic non-selective beta-blockers, growth hormone, non-routine vitamins or herbal products. Furthermore, thyroid hormones are not allowed unless the subject has used stable medication during the past 3 months.
59. Non-adherence to pre-dosing insulin regimen consisting of CSII
60. Subjects who meet one or more of dosing day exclusion criteria will be excluded from the dosing visit. In case a subject is excluded from the dosing visit, the dosing visit can be rescheduled 1-7 days later. Each of the dosing visits can only be rescheduled once.

    -

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Time in Range 70-180% | 24 hours
  Collection of clinical data regarding the treatment of two doses of 10mg dapagliflozin as add-on to night and day closed-loop control using the DreaMed Algorithm and the time within glucose range 70-180 mg/dl (3.9-10mmol/l) [%]

SECONDARY OUTCOMES:
urinary glucose excretion | 24 hours
  effect on urinary glucose excretion after a treatment with two doses of 10mg dapagliflozin (1x10 mg before bedtime and 1x10mg in the morning) in patients with type 1 diabetes
postprandial insulin need | 24 hours
  effect of postprandial insulin need after Treatment with dapagliflozin
ß-hydroxybutyrate | 24 hours
  association between Treatment of dapagliflozin and ß-hydroxybutyrate levels
Reduction of Insulin dose | 24 hours
  effect of insulin dose reduction during the DreaMed automated insulin delivery 24 hours after two doses of 10mg dapagliflozin in patients with type 1 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Danne, MD, Principal Investigator — Kinder- und Jugendkrankenhaus AUF DER BULT
Locations (1):
- Kinder - und Jugendkrankenhaus AUF DER BULT, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No